CLINICAL TRIAL: NCT00974701
Title: A Pilot and Feasibility Study to Evaluate Capsule Endoscopy in Subjects Presenting With Acute, Overt Upper Gastrointestinal Hemorrhage
Brief Title: A Pilot and Feasibility Study to Evaluate Capsule Endoscopy
Acronym: MA-79
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MA-79
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2010-05

CONDITIONS: Upper Gastrointestinal Hemorrhage
Keywords: symptoms of acute overt upper gastrointestinal hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients to undergo PillCam procedure (Experimental): Patients presenting to ER with acute overt upper GI bleeding
  Interventions: Device: PillCam ESO2

INTERVENTIONS:
Device: PillCam ESO2 — The capsule to be tested in this proposed study, PillCam ESO 2 capsule Endoscopy, is an improved version with exactly the same dimensions as the current PillCam ESO capsule, both in length and diameter.
  Other Names: PillCam ESO 2

SUMMARY:
This study is aimed at assessing the capability of the PillCam Platform using the PillCam ESO 2 Capsule in:

* Determining whether there is 1) active bleeding in the Upper gastrointestinal (UGI) tract, 2) identifying the anatomic location of acute overt UGI bleeding, and 3) discriminating a variceal versus non-variceal source of UGI bleeding.

DETAILED DESCRIPTION:
Upper gastrointestinal hemorrhage (UGIH) is a prevalent, clinically significant, and expensive healthcare problem worldwide. The incidence of acute, overt UGIH has been estimated to be 50-150 cases per 100,000 adults in the United States population each year.

Clinical Significance / Rationale EGD is the currently accepted community standard for the diagnosis and management of UGIH. Diagnostic EGD in persons presenting with acute UGIH allows for (1) differentiating the source of bleeding (variceal vs. non-variceal), (2) defining the anatomic location of the bleeding site (e.g., esophagus, stomach, duodenum), (3) providing an endoscopic diagnosis, and (4) facilitating patient triage for subsequent level of care (ICU, monitored bed, non-monitored bed, early / expedited hospital discharge).

Capsule endoscopy for the small bowel was cleared by the FDA in 2001, and within a short time, has gained acceptance as providing state-of-the-art endoscopic imaging. Capsule endoscopy is now commonly used in the evaluation of patients with obscure gastrointestinal bleeding, including iron deficiency anemia, suspected and known Crohn's disease, malabsorption syndromes (e.g., Celiac disease), and chronic abdominal pain. Capsule endoscopy technology is now also being applied to evaluation of the esophagus (PillCam® ESO, Given Imaging, Ltd, Yoqneam, Israel) and the colon (PillCam® COLON). Recently, a second generation esophageal capsule endoscope (PillCam® ESO 2, Given Imaging Ltd, Yoqneam, Israel) was cleared by the United States Food and Drug Administration in June 2007. While having the same outer dimensions (length and diameter) as the original PillCam ESO capsule, several significant improvements have been made to the internal components of the PillCam ESO 2. Similar to the original PillCam ESO, the system includes a sensor array and data recording device which are connected to the patient during the procedure. The recorded data is downloaded into the Given Imaging RAPID® workstation for review of the capsule endoscopy video.

However, there are no published detailed data evaluating the feasibility of utilizing PillCam ESO 2 in individuals presenting with acute, overt UGI bleeding. Moreover, there are no data comparing PillCam ESO 2 and EGD in the evaluation of this patient population. Therefore, in this proof-of-concept pilot study, we will evaluate the feasibility and safety of using PillCam ESO 2 in individuals presenting with acute, overt UGI bleeding.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* history of acute, overt UGI hemorrhage, defined as hematemesis (fresh blood or coffee grounds) and/or melena within the 48 hours prior to patient presentation

Exclusion Criteria:

* dysphagia
* odynophagia
* known swallowing disorder
* history of Zencker's diverticulum
* suspected bowel obstruction or bowel perforation at the time of presentation
* UGI hemorrhage with hemodynamic shock requiring urgent endoscopy
* history of prior bowel obstruction
* history of Crohn's disease
* history of UGI tract surgery (e.g., Billroth I, Billroth II, esophagectomy, gastrectomy, bariatric procedure)
* presence of an electromedical device (pacemaker or internal cardiac defibrillator)
* altered mental status (e.g., hepatic encephalopathy) at the time of presentation that would limit patient ability in swallowing the capsule
* pregnancy
* known allergy to conscious sedation medications
* known allergy to erythromycin
* inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Identification of gross blood (fresh or coffee grounds) / active bleeding in the esophagus, stomach and /or duodenum by PillCam™ ESO 2 and NG aspirate | 7 days

SECONDARY OUTCOMES:
Suspected anatomic location of acute overt UGI bleeding (e.g., esophageal, gastric, and/or duodenal location) by PillCam™ ESO 2 and EGD. | 7 days
Determination of suspected variceal vs. non-variceal source of acute overt UGIH by PillCam™ ESO 2 and EGD. | 7 days
Number, type and severity of adverse events and number of PillCam™ ESO 2 capsules that reached the 2nd portion of the duodenum. | 7 days
Patient subjective assessment questionnaires | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Josheph Sung, MD,PhD, Principal Investigator — Prince of Wales Hospital, Hong Kong, China; Ian Gralnek, MD., PhD., Principal Investigator — Rambam Medical Center, Haifa, Israel
Locations (2):
- Prince of Wales Hospital, Hong Kong, China, Shating, N.T., Hong Kong
- Rambma Medical Center, Haifa, Israel